CLINICAL TRIAL: NCT06064253
Title: Impact Of Health Education Program on Adherence to Treatment in Egyptian Patients With Knee Osteoarthritis
Brief Title: Adherence to Treatment in Egyptian Patients With Knee Osteoarthritis
Acronym: OA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Amany Mohammed Ibrahim Ebaid, Associate professor, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB #:4677
Record Dates: First submitted 2023-09-24; First posted 2023-10-03 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Knee Osteoarthritis
Keywords: Osteoarthritis; Knee; Adherence; Patient education; Guidelines
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Other): health education program explaining the nature of the condition(KOA causes, pathological changes, and natural course of the disease), we explained the recommendations for the treatment of KOA, teaching the patient a home exercise program of 5 exercises (targeting knee extensor and hip muscle ), selection of a physiotherapy program suitable to the patient clinical condition, recommendations to increase daily physical activity ( e.g. brisk walking) with joint protection measures along with a weight reduction regimen proposed in overweight and obese patients and prescribing a suitable pharmacological treatment to the patients
  Interventions: Behavioral: health education
- control group (No Intervention): were assigned the traditional approach for KOA management, they were told their diagnosis if they were not already familiar with it, received the treatment for KOA according to ACR guidelines, they were offered physical therapy modalities if their condition required but they were not given the health education program or the other interventional steps.

INTERVENTIONS:
Behavioral: health education — adherence to treatment
  Other Names: exercise and diet plan
  Arms: intervention group

SUMMARY:
the aim is to measure the level of adherence of knee osteoartheritis patients to a Carefully curated program that follows the American College of Rheumatology/Arthritis (ACR) recommendation guidelines and investigate the factor that might affect the patient's adherence to the prescribed protocol.

DETAILED DESCRIPTION:
2.3. interventional protocol (for intervention group only): For the Intervention group: A face-to-face semi-structured interview was carried out with each participant separately. The interview (30-45minuts) included a health education program explaining the nature of the condition(KOA causes, pathological changes, and natural course of the disease), we explained the recommendations for the treatment of KOA, teaching the patient a home exercise program of 5 exercises (targeting knee extensor and hip muscle ), selection of a physiotherapy program suitable to the patient clinical condition, recommendations to increase daily physical activity ( e.g. brisk walking) with joint protection measures along with a weight reduction regimen proposed in overweight and obese patients and prescribing a suitable pharmacological treatment to the patients mentioning side effect that might occur. At the end of the interview, each participant received a booklet including the recommendations for the treatment of knee osteoarthritis according to the ACR.

As for the control group, they were assigned the traditional approach for KOA management, they were told their diagnosis if they were not already familiar with it, received the treatment for KOA according to ACR guidelines, they were offered physical therapy modalities if their condition required but they were not given the health education program or the other interventional steps.

2.4. Follow-up period: Throughout the following three months after enrollment, participants were followed up every ten days; asking about persistence on the prescribed treatment and exercise program, the level of their daily activity, and their diet plan. For participants who failed to attend for any reason, a telephone call was performed to provide behavior change support in both groups. The telephone call aimed to observe adherence to treatment in the control group and to increase levels of participation in the intervention group.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed as having knee osteoarthritis according to the American College of Rheumatology criteria

Exclusion Criteria:

* Patients with a

  1. A history of knee trauma or injury
  2. patients suffering from any other rheumatological diseases (e.g., Rheumatoid Arthritis)
  3. severe comorbidities, severe cardiovascular disease, heart failure, gastrointestinal bleeding risk, and chronic kidney disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2023-01-12 (Actual); Primary Completion 2023-05-24 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
measuring KOA patients adherence | 3 months
  adherence survey based on morsiky adherence scale
improved patients function and improved patient pain | 3 MONTHS
  measured by Western Ontario and McMaster University Osteoarthritis Index contains 5 items that address the following person-level activities: walking, stair climbing, sitting, lying down, and standing
  --measured by visual analog scale

SECONDARY OUTCOMES:
investigating the factors that hinder patient adherence | 3 months
  WHO frame work foe adherence

CONTACTS AND LOCATIONS:
Locations (1):
- Zagazig University Hospitals, Zagazig, Sharqia Province, Egypt